CLINICAL TRIAL: NCT02425475
Title: A Prospective, Non-controlled, Multicenter Clinical Study to Evaluate the Diagnostic Accuracy of the Stepwise Two Photon Excited Melanin Fluorescence of Potentially Malignant Pigmented Lesions as Compared to Histopathological Diagnosis
Brief Title: FLuorescence Identification of Melanoma by a Multicenter Based Algorithm (FLIMMA)
Acronym: FLIMMA
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Heidelberg (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: FLIMMA-01
Record Dates: First submitted 2015-04-02; First posted 2015-04-24 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Melanoma; Moles
Keywords: Dermoscopy
MeSH Terms: conditions — Melanoma; Nevus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mole: Patients with suspicious moles
  Interventions: Device: LIMES

INTERVENTIONS:
Device: LIMES — All patients will undergo dermoscopic diagnosis and be documented with a video image storing. The diagnosis based on dermoscopy will be immediately documented. Then, as a second diagnostic procedure, fluorescence diagnostics based on the two photon excitation from a dye-laser will be performed. The classification as non-melanoma or malignant melanoma by the medical device LIMES will also be documented immediately. Afterwards, the lesion will be excised and undergo histo-pathologic examination by the respective histopathologist of the participating centers. The histopathologic diagnosis will serve as gold standard for subsequent evaluations of the diagnostic accuracy.

SUMMARY:
All patients will undergo dermoscopic diagnosis and be documented with a video image storing. The diagnosis based on dermoscopy will be immediately documented. Then, as a second diagnostic procedure, fluorescence diagnostics based on the two photon excitation from a dye-laser will be performed. The classification as non-melanoma or malignant melanoma by the medical device LIMES will also be documented immediately. Afterwards, the lesion will be excised and undergo histopathologic examination by the respective histopathologist of the participating centers. The histopathologic diagnosis will serve as gold standard for subsequent evaluations of the diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Male or female
* Patients having pigmented lesions with suspicion of dysplastic nevus or melanoma, in whom an excision is performed in order to exclude or diagnose malignant melanoma
* Patients who gave their written informed consent.

Exclusion Criteria:

* Patients with skin type V and VI according to Fitzpatrick's scale;
* Where there is a risk that the scanning head is torn off be-cause the patient cannot be placed at rest (e.g. due to motoric disorders like tremor, convulsions, tics, compulsive acts
* Patients who cannot understand the patient information and provide informed consent
* Deep dermal lesions ≥ 5 mm beneath the stratum corneum
* Clinically or reflected-light microscopically obviously non-melanocytic lesions
* Peri- and subungual lesions
* Mucosal lesions
* Lesions with trauma, erosion (superficial defect), excoriation (defect down to the basement membrane) or ulceration (deep substantial defect) on more than 50 % of the lesion area (measurements must in any case not be carried out directly on the trauma, erosion, excoriation or ulceration)
* Tattooed lesions
* Pregnant or breast feeding women
* Patients suffering from albinism
* Lesions with dominant (>50%) regression
* Lesions which are not suitable to fix the scanning cap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study evaluates patients with pigmented lesions, which are excised in order to exclude or diagnose cutaneous melanoma.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To determine sensitivity and specificity of the algorithm for the fluorescence diagnostics of melanoma. | 7 days
  The comparator and gold standard for the diagnosis will be the histopathological diagnosis of the pigmented lesions.

SECONDARY OUTCOMES:
To collect data for training and optimization of the diagnostic algorithm. | 1 day

OTHER OUTCOMES:
To assess the safety of the device and to assess the incidence of adverse events | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, MD, Principal Investigator — Dept. of Dermatology, University Hospital Tübingen
Locations (3):
- Germany (3):
  - Dept. of Dermatology, Charité, Berlin
  - Dept. of Dermatology, University Hospital, Heidelberg
  - Dept. of Dermatology, University Hospital, Tübingen

REFERENCES:
- [Derived] Hofmann MA, Keim U, Jagoda A, Forschner A, Fink C, Spankuch I, Tampouri I, Eigentler T, Weide B, Haenssle HA, Garbe C. Dermatofluoroscopy diagnostics in different pigmented skin lesions: Strengths and weaknesses. J Dtsch Dermatol Ges. 2020 Jul;18(7):682-690. doi: 10.1111/ddg.14163. Epub 2020 Jul 12. PMID 32657017
- [Derived] Fink C, Hofmann M, Jagoda A, Spaenkuch I, Forschner A, Tampouri I, Lomberg D, Leupold D, Garbe C, Haenssle HA. Study protocol for a prospective, non-controlled, multicentre clinical study to evaluate the diagnostic accuracy of a stepwise two-photon excited melanin fluorescence in pigmented lesions suspicious for melanoma (FLIMMA study). BMJ Open. 2016 Dec 19;6(12):e012730. doi: 10.1136/bmjopen-2016-012730. PMID 27993903